CLINICAL TRIAL: NCT04236141
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Polatuzumab Vedotin in Combination With Bendamustine and Rituximab Compared With Bendamustine and Rituximab Alone in Chinese Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma.
Brief Title: A Study to Evaluate the Efficacy and Safety of Polatuzumab Vedotin in Combination With Bendamustine and Rituximab Compared With Bendamustine and Rituximab Alone in Chinese Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL).
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision, no safety concerns
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YO41543
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Polatuzumab Vedotin plus BR (Experimental)
  Interventions: Drug: Polatuzumab Vedotin; Drug: Bendamustine; Drug: Rituximab
- Placebo plus BR (Active Comparator)
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Participants will receive a total of 6 cycles (a cycle being 21 days) of 1.8mg/kg Polatuzumab Vedotin (IV infusion) on Day 2 of Cycle 1 and Day 1 of Cycles 2-6.
  Arms: Polatuzumab Vedotin plus BR
Drug: Bendamustine — Participants will receive a total of 6 cycles (a cycle being 21 days) of 90 mg/m2 Bendamustine (IV infusion) on Days 2 and 3 of Cycle 1 and Days 1 and 2 of Cycles 2-6.
Drug: Rituximab — Participants will receive a total of 6 cycles (a cycle being 21 days) of 375 mg/m2 Rituximab (IV infusion) on Day 1 of each cycle.
Drug: Placebo — Participants will receive a total of 6 cycles (a cycle being 21 days) of Placebo (IV infusion) on Day 2 of Cycle 1 and Day 1 of Cycles 2-6.
  Arms: Placebo plus BR

SUMMARY:
A study to evaluate the Efficacy and Safety of Polatuzumab Vedotin in combination with BR (Bendamustine and Rituximab) compared with BR alone in Chinese participants with R/R DLBCL. Approximately 42 Chinese participants will be randomised to treatment arms in a 2:1 ratio. Randomisation will be conducted with the aid of an interactive web-based response system (IxRS).

ELIGIBILITY:
Inclusion Criteria:

* Able to comply with the study protocol and procedures, in the investigator's judgement.
* Transplant ineligible participants with R/R DLBCL.
* Confirmed DLBCL diagnosis.
* For participants who have received prior bendamustine, a response duration > 1 year (for participants who have relapsed disease after a prior regimen).
* At least one bi-dimensionally measurable lesion, defined as > 1.5 cm in its longest dimension as measured by CT or magnetic resonance imaging (MRI).
* Availability of archival or freshly collected tumor tissue before study enrolment.
* Life expectancy of at least 24 weeks.
* ECOG Performance Status of 0, 1 or 2.
* Adequate haematologic function.
* Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs.
* For men who are not surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating sperm.
* Residence in the People's Republic of China.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (MAbs) or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products.
* Contraindication to bendamustine or rituximab.
* History of sensitivity to mannitol (mannitol is an excipient in bendamustine).
* Prior use of any MAb, radioimmunoconjugate, or antibody-drug conjugate (ADC) within 5 half-lives or 4 weeks, whichever is longer, before Cycle 1, Day 1.
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to Cycle 1, Day 1.
* Ongoing corticosteroid use > 30 mg/day prednisone or equivalent, for purposes other than lymphoma symptom control.
* Completion of autologous SCT within 100 days prior to Cycle 1, Day 1.
* Prior allogeneic Stem Cell Transplantation (SCT).
* Prior treatment with Chimeric Antigen Receptor (CAR) T-cell therapy.
* Eligibility for autologous SCT.
* Grade 3b Follicular Lymphoma (FL).
* History of transformation of indolent disease to DLBCL.
* Primary or secondary CNS lymphoma.
* Current Grade > 1 peripheral neuropathy.
* History of other malignancy that could affect compliance with the protocol or interpretation of results.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular or pulmonary disease.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1.
* Participants with suspected or latent tuberculosis.
* Positive Chronic Hepatitis B (HBV) infection or Hepatitis C (HCV) infection.
* Known history of HIV infection.
* Known infection human T-cell leukemia virus 1 virus.
* Vaccination with a live vaccine within 28 days prior to treatment.
* Recent major surgery (within 6 weeks before the start of Cycle 1, Day 1) other than for diagnosis.
* Pregnant or breastfeeding or intending to become pregnant during the study or within 12 months after the final dose of study treatment.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- China (10):
  - Beijing Cancer Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in mainland China from 10 July 2020 to 07 February 2022.
Pre-assignment Details: A total of 42 participants were randomized in the study with a randomization ratio 2:1. Of the 42 participants randomized, 41 participants received at least one dose of study drug and their intended treatment.
Groups:
- Polatuzumab Vedotin Plus Bendamustine and Rituximab: Participants received polatuzumab vedotin administered at an initial dose of 1.8 milligrams per kilogram (mg/kg), as intravenous (IV) infusion on Day 2 of Cycle 1 and thereafter on Day 1 of Cycles 2-6.
  Participants also received bendamustine, 90 milligrams per square meter (mg/m^2), as IV infusion, on Days 2 and 3 of Cycle 1 and thereafter on Days 1 and 2 of Cycles 2-6 and rituximab, 375 mg/m^2, as IV infusion, at least 30 minutes before the administration of other study treatments, on Day 1 of Cycles 1-6, concurrently with polatuzumab vedotin. Each cycle is 21 days.
- Placebo Plus Bendamustine and Rituximab: Participants received polatuzumab vedotin matching placebo by IV infusion on Day 2 of Cycle 1 and thereafter on Day 1 of Cycles 2-6.
  Participants also received bendamustine, 90 mg/m^2, as IV infusion, on Days 2 and 3 of Cycle 1 and thereafter on Days 1 and 2 of Cycles 2-6 and rituximab, 375 mg/m^2, as IV infusion, at least 30 minutes before the administration of other study treatments, on Day 1 of Cycles 1-6, concurrently with placebo. Each cycle is 21 days.
Period: Overall Study
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Started | 28 | 14
Safety Population (Safety population included all randomized participants who received at least one dose of the study drug.) | 27 | 14
Pharmacokinetic-Evaluable Population (Pharmacokinetic (PK)-evaluable population included all participants who had at least one evaluable PK sample post dose for at least one analyte.) | 27 | 0
Immunogenicity-Evaluable Population (Baseline Evaluable) (Immunogenicity-evaluable population included all participants with anti-drug antibody (ADA) assay results from baseline sample.) | 27 | 14
Immunogenicity-Evaluable Population (Post-Baseline Evaluable) (Immunogenicity-evaluable population included all participants with at least one evaluable post-baseline ADA sample) | 24 | 0
Intent-to-treat Population (Intention-to-treat (ITT) population included all participants randomized, whether or not the participants received the assigned treatment.) | 28 | 14
Completed | 0 | 0
Not Completed | 28 | 14
Not completed — Death | 18 | 10
Not completed — Withdrawal by Participant | 1 | 0
Not completed — Reason not Specified | 1 | 0
Not completed — Study terminated by Sponsor | 8 | 4

BASELINE CHARACTERISTICS:
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Groups:
- Polatuzumab Vedotin Plus Bendamustine and Rituximab: Participants received polatuzumab vedotin administered at an initial dose of 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 and thereafter on Day 1 of Cycles 2-6.
  Participants also received bendamustine, 90 mg/m^2, as IV infusion, on Days 2 and 3 of Cycle 1 and thereafter on Days 1 and 2 of Cycles 2-6 and rituximab, 375 mg/m^2, as IV infusion, at least 30 minutes before the administration of other study treatments, on Day 1 of Cycles 1-6, concurrently with polatuzumab vedotin. Each cycle is 21 days.
- Total: Total of all reporting groups
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Continuous [Median (Full Range); unit: years] | 57.00 [27.0 to 70.0] | 60.50 [31.0 to 76.0] | 58.00 [27.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 21 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 14 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 14 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) at the End of Treatment (EOT) Assessment Based on Positron Emission Tomography-Computed Tomography (PET-CT) Assessed by Independent Review Committee (IRC)
Description: CR was determined by IRC according to the Lugano Response Criteria (LRC) for Malignant Lymphoma. Per LRC , CR based on PET-CT was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS), where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 25.0 [10.69 to 44.87] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 10.71, 95% CI 2-sided [-19.00 to 40.43]

2. Secondary Outcome: Percentage of Participants With CR at the EOT Assessment Based on PET-CT as Assessed by Investigator
Description: CR was determined by investigator according to the LRC for Malignant Lymphoma. Per LRC, CR based on PET-CT was defined as complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5PS, where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment. Percentages have been rounded off to the first decimal point.
Time Frame: Up to approximately to 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 21.4 [8.30 to 40.95] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 7.14, 95% CI 2-sided [-22.03 to 36.31]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR) at EOT Based on PET-CT as Assessed by Investigator
Description: OR was defined as CR or partial response (PR) at the end of treatment assessment based on PET-CT, as determined by the investigator according to the LRC. CR based on PET-CT was defined as complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass on 5PS, where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. PR based on PET-CT was defined as partial MR in lymph nodes and extralymphatic sites with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size; no new lesions and residual uptake higher than uptake in normal bone marrow but reduced compared with baseline. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 28.6 [13.22 to 48.67] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 14.29, 95% CI 2-sided [-15.89 to 44.46]

4. Secondary Outcome: Percentage of Participants With OR at EOT Based on PET-CT as Assessed by IRC
Description: OR was defined as CR or PR at the end of treatment assessment based on PET-CT, as determined by the IRC according to the LRC. CR based on PET-CT was defined as complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass on 5PS, where, 1= no uptake above background; 2 = uptake ≤ mediastinum; 3 = uptake > mediastinum but ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. PR per PET-CT was defined as partial MR in lymph nodes and extralymphatic sites with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size; no new lesions and residual uptake higher than uptake in normal marrow but reduced compared with baseline. The analysis was done 6-8 weeks after Cycle 6, Day 1(1 cycle= 21 days) or after final dose of study treatment.Percentages have been rounded off to the first decimal point.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 35.7 [18.64 to 55.93] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 21.43, 95% CI 2-sided [-9.44 to 52.30]

5. Secondary Outcome: Percentage of Participants With CR at EOT Based on Computed Tomography (CT) as Assessed by Investigator
Description: CR was determined by the investigator according to the LRC. Per LRC, CR based on CT was defined as complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 centimeters (cm) in longest transverse diameter (LDi) and no extralymphatic sites of disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, immunohistochemistry (IHC) negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 17.9 [6.06 to 36.89] | 0 [0.00 to 23.16]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 17.86, 95% CI 2-sided [-1.69 to 37.40]

6. Secondary Outcome: Percentage of Participants With CR at EOT Based on CT as Assessed by IRC
Description: CR was determined by the IRC according to the LRC. Per LRC, CR based on CT was defined as complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no extralymphatic sites of disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 17.9 [6.06 to 36.89] | 0 [0.00 to 23.16]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 17.86, 95% CI 2-sided [-1.69 to 37.40]

7. Secondary Outcome: Percentage of Participants With OR at EOT Assessment Based on CT as Assessed by Investigator
Description: OR was defined as CR or PR, at the EOT assessment based on CT only, as determined by the investigator according to the LRC. Per LRC, CR based on CT was defined as complete radiologic response in lymph nodes and extralymphatic sites with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no extralymphatic sites of disease; absence of non-measured lesion; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. Per LRC, PR was defined as ≥ 50% decrease in sum of the product of the perpendicular diameters (SPD) of up to 6 target nodes and extranodal sites; non-measured lesion is absent/normal, regressed, but no increase; spleen must have regressed by >50 % in length beyond normal; and no new lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment. Percentages have been rounded off to the first decimal point.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 32.1 [15.88 to 52.35] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 17.86, 95% CI 2-sided [-12.70 to 48.42]

8. Secondary Outcome: Percentage of Participants With OR at EOT Assessment Based on CT as Assessed by IRC
Description: OR was defined as percentage of participants with CR or PR, at EOT assessment based on CT only, as determined by IRC according to the LRC. Per LRC, CR based on CT was defined as complete radiologic response with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi. PR is ≥ 50% decrease in SPD of up to 6 target nodes and extranodal sites. The analysis was done 6-8 weeks after Cycle 6, Day 1 (1 cycle = 21 days) or after final dose of study treatment.
Time Frame: Up to approximately 23 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 28.6 [13.22 to 48.67] | 14.3 [1.78 to 42.81]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 14.29, 95% CI 2-sided [-15.89 to 44.46]

9. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) Based on PET-CT or CT Only as Assessed by Investigator
Description: BOR=CR/PR per PET-CT/CT by investigator per LRC.CR perPET-CT=complete MR in lymph nodes & extralymphatic sites(ELS),score=1,2,3 with/without residual mass on5PS,1=no uptake(UT)above background;2=UT≤mediastinum;3=UT>mediastinum but ≤liver;4=UT moderately>liver;5=UT markedly higher than liver and/or new lesions; no new lesions & FDG-avid disease absent in bone marrow.CR perCT=complete radiologic response with target nodes/nodal masses regressedto≤1.5 cm in LDi&no ELS of disease;absence of non-measured lesion;organ enlargement regressed to normal;no new lesions;bone marrow morphology=normal,if indeterminate,IHC negative.PR per PET-CT=partial MR in lymph nodes&ELS,score=4or5,reduced UT than baseline(BL)&residual masses=any size;no new lesions&residual UT >UT in normal marrow,reduced than BL.PR per CT by LCR=≥50% decrease in SPD of up to 6 target nodes & extranodal sites;non-measured lesion=absent/normal,regressed,no increase;spleen=regressed by>50%in length beyond normal;no new lesions.
Time Frame: Up to every 6 months after end of treatment assessment until disease progression, study withdrawal, end of study, or death, whichever occurred first (up to approximately 82 weeks)
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 53.6 [33.87 to 72.49] | 28.6 [8.39 to 58.10]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 25.00, 95% CI 2-sided [-10.38 to 60.38]

10. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) Based on PET-CT or CT Only as Assessed by IRC
Description: BOR=CR/PR per PET-CT/CT by IRC per LRC. CR per PET-CT=complete MR in lymph nodes& ELS, score=1, 2,3 with/without residual mass on 5PS, 1=no UT above background; 2=UT≤mediastinum; 3=UT>mediastinum but ≤liver; 4=UT moderately>liver; 5=UT markedly higher than liver and/or new lesions; no new lesions & FDG-avid disease absent in bone marrow.CR per CT=complete radiologic response with target nodes/nodal masses regressed to≤1.5 cm in LDi and no ELS of disease; absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; bone marrow morphology=normal, if indeterminate, IHC negative. PR per PET-CT=partial MR in lymph nodes & ELS, score =4 or 5,reduced UT than baseline(BL)&residual masses=any size; no new lesions &residual UT >UT in normal marrow, reduced than BL.PR per CT by LCR=≥50% decrease in SPD of up to 6 target nodes& extranodal sites; non-measured lesion=absent/normal, regressed, no increase; spleen=regressed by>50% in length beyond normal; no new lesions.
Time Frame: as for outcome 9
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
percentage of participants | 53.6 [33.87 to 72.49] | 50.0 [23.04 to 76.96]
Statistical Analysis 1: Comparison: Polatuzumab Vedotin Plus Bendamustine and Rituximab vs Placebo Plus Bendamustine and Rituximab; Test type: Superiority; Difference in Response Rates = 3.57, 95% CI 2-sided [-33.84 to 40.98]

11. Secondary Outcome: Duration Of Response (DOR) Based on PET-CT/CT Only as Assessed by Investigator
Description: DOR was defined as time from first occurrence of a documented objective response to disease progression, relapse or death from any cause, as determined by the investigator according to the LRC
Time Frame: as for outcome 9
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment. Overall number of participants analyzed are the number of BOR responders as assessed by investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 15 | 4
months | 5.45 [3.91 to 8.67] | 4.34 [2.60 to NA] — The upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events.

12. Secondary Outcome: DOR Based on PET-CT/CT Only as Assessed by IRC
Description: DOR was defined as time from first occurrence of a documented objective response to disease progression, relapse or death from any cause, as determined by IRC according to the LRC.
Time Frame: as for outcome 9
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment. Overall number of participants analyzed are the number of BOR responders assessed by IRC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 15 | 7
months | 8.74 [3.55 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events. | 4.27 [2.60 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events.

13. Secondary Outcome: Progression-Free Survival (PFS) Based on PET-CT/CT Only as Assessed by Investigator
Description: PFS was defined as the period from date of randomization until the date of disease progression, relapse, or death from any cause based on PET-CT or CT only, as determined by the investigator according to the LRC.
Time Frame: Up to approximately 82 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
months | 4.90 [3.12 to 6.60] | 2.00 [1.87 to 4.60]

14. Secondary Outcome: PFS Based on PET-CT/CT Only as Assessed by IRC
Description: PFS was defined as the period from date of randomization until the date of disease progression, relapse, or death from any cause based on PET-CT or CT only, as determined by IRC according to the LRC.
Time Frame: Up to approximately 82 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
months | 5.42 [4.47 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events. | 6.01 [3.52 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events.

15. Secondary Outcome: Event-Free Survival (EFS) Based on PET-CT or CT Assessed by Investigator
Description: EFS was defined as the time from date of randomization to any treatment failure including disease progression, relapse, initiation of new anti-lymphoma treatment (NALT), or death based on PET-CT or CT only, as determined by the investigator according to the LRC.
Time Frame: Up to approximately 82 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
months | 4.83 [3.12 to 6.44] | 2.00 [1.87 to 4.60]

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization until the date of death from any cause.
Time Frame: Up to approximately 82 weeks
Population: ITT population included all participants randomized, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 28 | 14
months | 10.89 [5.52 to 16.66] | 7.67 [6.01 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events.

17. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An adverse event can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), recurrence of an intermittent medical condition not present at baseline, any deterioration in a laboratory value or other clinical test that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug or adverse events that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment.
Time Frame: Up to approximately 82 weeks
Population: Safety population included all randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
Number analyzed (Participants) | 27 | 14
percentage of participants | 100 | 100

18. Secondary Outcome: Serum Concentration of Total Antibody at Specified Timepoints
Description: PK of polatuzumab vedodtin-related analyte- total antibody was measured
Time Frame: Predose & post dose on Day 2 of Cycle 1,& post dose on Days 8 & 15 of Cycles 1& 3; predose & post dose on Day 1 of Cycles 2, 3 & 4; treatment completion/early discontinuation visit; follow-up visits at Months 3 &6 (1 cycle=21 days) up to approx. 46 weeks
Population: PK-evaluable population included all participants who had at least one evaluable PK sample post dose for at least one analyte. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab
Number analyzed (Participants) | 27
micrograms per milliliter (μg/mL)
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as all samples were below the limit of quantification (BLQ).
  Cycle 1 Day 2: Post dose | 41.5 (26.3)
  Cycle 1 Day 8 Post dose: number analyzed (Participants) | 23
  Cycle 1 Day 8 Post dose | 9.83 (38.3)
  Cycle 1 Day 15 Post dose: number analyzed (Participants) | 26
  Cycle 1 Day 15 Post dose | 5.42 (35.6)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 24
  Cycle 2 Day 1: Pre-dose | 3.13 (37.3)
  Cycle 2 Day 1: Post dose: number analyzed (Participants) | 24
  Cycle 2 Day 1: Post dose | 49.1 (39.6)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Pre-dose | 4.30 (36.3)
  Cycle 3 Day 1: Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Post dose | 45.6 (28.9)
  Cycle 3 Day 8 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 8 Post dose | 13.6 (29.1)
  Cycle 3 Day 15 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 15 Post dose | 8.48 (30.8)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Pre-dose | 5.37 (52.5)
  Cycle 4 Day 1: Post dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Post dose | 47.2 (34.8)
  Treatment completion/Early discontinuation: number analyzed (Participants) | 22
  Treatment completion/Early discontinuation | 4.44 (49.5)
  Follow-Up Month 3: number analyzed (Participants) | 8
  Follow-Up Month 3 | 0.182 (NA) — Since more than one-third values were BLQ, the geometric coefficient of variation was not estimable.
  Follow-Up Month 6: number analyzed (Participants) | 3
  Follow-Up Month 6 | 0.0410 (NA) — Since more than one-third values were BLQ, the geometric coefficient of variation was not estimable.

19. Secondary Outcome: Plasma Concentration of Antibody-Conjugated Monomethyl Auristatin E (acMMAE) at Specified Timepoints
Description: PK of polatuzumab vedodtin-related analyte- acMMAE was measured.
Time Frame: Predose and post dose on Day 2 of Cycle 1, and post dose on Days 8 and 15 of Cycles 1 and 3; predose and post dose on Day 1 of Cycles 2, 3 and 4; treatment completion/early discontinuation visit (each cycle = 21 days) up to approximately 19 weeks
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab
Number analyzed (Participants) | 27
nanograms per milliliter (ng/mL)
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as all samples were BLQ.
  Cycle 1 Day 2: Post dose | 560 (23.0)
  Cycle 1 Day 8 Post dose: number analyzed (Participants) | 24
  Cycle 1 Day 8 Post dose | 65.5 (212.3)
  Cycle 1 Day 15 Post dose: number analyzed (Participants) | 26
  Cycle 1 Day 15 Post dose | 26.7 (35.7)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 23
  Cycle 2 Day 1: Pre-dose | 10.9 (35.9)
  Cycle 2 Day 1: Post dose: number analyzed (Participants) | 24
  Cycle 2 Day 1: Post dose | 524 (97.4)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Pre-dose | 14.6 (36.1)
  Cycle 3 Day 1: Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Post dose | 605 (19.5)
  Cycle 3 Day 8 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 8 Post dose | 64.5 (210.3)
  Cycle 3 Day 15 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 15 Post dose | 33.7 (31.7)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Pre-dose | 15.4 (56.2)
  Cycle 4 Day 1: Post dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Post dose | 602 (19.4)
  Treatment completion/Early discontinuation: number analyzed (Participants) | 22
  Treatment completion/Early discontinuation | 10.6 (49.1)

20. Secondary Outcome: Plasma Concentration of Unconjugated Monomethyl Auristatin E (MMAE) at Specified Timepoints
Description: PK of polatuzumab vedodtin-related analyte- unconjugated MMAE was measured.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab
Number analyzed (Participants) | 27
ng/mL
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as all samples were BLQ.
  Cycle 1 Day 2: Post dose | 0.139 (81.9)
  Cycle 1 Day 8 Post dose: number analyzed (Participants) | 23
  Cycle 1 Day 8 Post dose | 2.47 (50.6)
  Cycle 1 Day 15 Post dose: number analyzed (Participants) | 26
  Cycle 1 Day 15 Post dose | 0.627 (64.1)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 24
  Cycle 2 Day 1: Pre-dose | 0.0870 (106.8)
  Cycle 2 Day 1: Post dose: number analyzed (Participants) | 24
  Cycle 2 Day 1: Post dose | 0.127 (72.2)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Pre-dose | 0.0944 (65.9)
  Cycle 3 Day 1: Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 1: Post dose | 0.171 (44.1)
  Cycle 3 Day 8 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 8 Post dose | 1.49 (149.6)
  Cycle 3 Day 15 Post dose: number analyzed (Participants) | 23
  Cycle 3 Day 15 Post dose | 0.509 (58.7)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Pre-dose | 0.0851 (130.9)
  Cycle 4 Day 1: Post dose: number analyzed (Participants) | 18
  Cycle 4 Day 1: Post dose | 0.152 (64.6)
  Treatment completion/Early discontinuation: number analyzed (Participants) | 22
  Treatment completion/Early discontinuation | 0.0711 (98.0)

21. Secondary Outcome: Number of Participants With Positive Treatment Emergent Anti-Drug Antibodies (ADA) to Polatuzumab Vedotin
Description: Treatment Emergent ADA is (a) negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result, OR (b) positive ADA result at baseline and one or more post-baseline titer results that are at least 0.60 titer unit (t.u.) greater than the baseline titer result.
Time Frame: Baseline up to approximately 39 weeks
Population: Immunogenicity-evaluable population (Post-Baseline Evaluable) included all participants with at least one evaluable post-baseline anti-drug antibody (ADA) sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 82 weeks
Description: All-cause mortality is reported for all enrolled participants. Serious and other adverse events are reported for safety population which included all participants who received at least 1 dose of study drug.
Arm/Group | Polatuzumab Vedotin Plus Bendamustine and Rituximab | Placebo Plus Bendamustine and Rituximab
All-Cause Mortality (participants affected / at risk) | 18/28 | 10/14
Serious Adverse Events (participants affected / at risk) | 12/27 | 3/14
Other Adverse Events (participants affected / at risk) | 27/27 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polatuzumab Vedotin Plus Bendamustine and Rituximab (N=27) | Placebo Plus Bendamustine and Rituximab (N=14)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polatuzumab Vedotin Plus Bendamustine and Rituximab (N=27) | Placebo Plus Bendamustine and Rituximab (N=14)
Anaemia (Blood and lymphatic system disorders) | 16 (28) | 5 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (11) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (21) | 4 (7)
Vomiting (Gastrointestinal disorders) | 10 (19) | 4 (5)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 9 (13) | 5 (5)
Malaise (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 10 (15) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (13) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (13) | 1 (3)
Bilirubin conjugated increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 5 (7) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 5 (5) | 0 (0)
Blood potassium decreased (Investigations) | 2 (3) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 2 (3) | 0 (0)
C-reactive protein increased (Investigations) | 3 (3) | 0 (0)
Electrocardiogram high voltage (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (4) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (13) | 10 (16)
Lymphocyte percentage decreased (Investigations) | 1 (2) | 1 (1)
Mononuclear cell count increased (Investigations) | 1 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 19 (51) | 7 (18)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0)
Neutrophil percentage increased (Investigations) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 15 (24) | 7 (9)
Protein urine present (Investigations) | 2 (2) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 1 (1)
White blood cell count decreased (Investigations) | 20 (56) | 9 (20)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (23) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Venous thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT04236141/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04236141/SAP_001.pdf